CLINICAL TRIAL: NCT07024914
Title: Effect of Oxygen Supplementation on Cerebral Oxygenation, Symptoms and Performance During 30 Sec STST in Chronic Obstructivepulmonary Disease Patients, Without Resting Hypoxemia
Brief Title: Effect of Oxygen Supplementation on Cerebral Oxygenation, Symptoms and Performance During STST in COPD Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Afroditi Boutou, Consultant in Pulmonary Medicine, George Papanicolaou Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GeorgePH39/16-01-2019
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation of oxygen during the 30 sec Sit to Stand Test in patients with COPD (Active Comparator): Oxygen supplementation via nasal cannula at a rate of 3 lit/min
  Interventions: Drug: Oxygen
- Supplementation of medical air during the 30 sec Sit to Stand Test in patients with COPD (Sham Comparator): Medical air supplementation via nasal cannula at a rate of 3 lit/min
  Interventions: Drug: medical air

INTERVENTIONS:
Drug: Oxygen — Oxygen supplementation via nasal cannula at a rate of 3 lit/min during 30sec Sit-To-Stand Test among COPD patients without resting hypoxemia
  Arms: Supplementation of oxygen during the 30 sec Sit to Stand Test in patients with COPD
Drug: medical air — Medical Air supplementation via nasal cannula at a rate of 3 lit/min during 30sec Sit-To-Stand Test among COPD patients without resting hypoxemia
  Arms: Supplementation of medical air during the 30 sec Sit to Stand Test in patients with COPD

SUMMARY:
It is a randomised, single-blind trial of the effect of acute oxygen supplementation on cerebral oxygenation during the 30 sec Sit-To-Stand Test (STST) in chronic obstructive pulmonary disease patients, without resting hypoxemia. After an initial clinical assessment, patients preform the 30sec STST under near-infrared spectroscopy, a non invasive technique which assesses cerebral oxygenation at the prefrontal lobe. Measurements are performed twice, under oxygen supplementation or medical air, in a random order, and the patients are be blinded to the treatment (oxygen or medical air) given.

ELIGIBILITY:
Inclusion Criteria:

1) clinical diagnosis of COPD, based on smoking history of at least 100 cigarettes and post bronchodilation forced expiratory volume (FEV1) to forced vital capacity (FVC) ratio <0.7, and 2) resting arterial oxygen partial pressure >60 mmHg, according to recent (within a week) arterial blood gases assessment.

Exclusion Criteria:

1) recent COPD exacerbation (as indicated by deterioration of respiratory symptoms, hospital admission and/or change in medication within the previous month), 2) history of specific balance problems (i.e., diagnosed neurological or vestibular disorder), 3) spinal surgery, and 4) lower limb musculoskeletal problems (i.e., surgery, injury or pathology at hip, knee, ankle or foot)

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
cerebral oxygenation at the prefrontal lobe | For 2 and a half minutes (one minute of rest, 30 seconds during Sit-To-Stand Test and one minute of recovery after the test)
  Near infrared spectroscopy will be utilised to assess cerebral oxygenation, by measuring oxygenated hemoglobin (O2Hb) at the prefrontal lobe, in COPD patients

SECONDARY OUTCOMES:
Number of repetitions during Sit-To-Stand Test | From the initiation till the end of the Sit-To-Stand Test, that is 30 seconds.
  The number of repetitions (fully standing and sitting) during the Sit-To-Stand Test
Severity of dyspnea | At the end of the 30 second Sit-To-Stand Test
  Rate of dyspnea according to dyspnea Borg scale (0-10)
Severity of fatigue | At the end of the 30 seconds Sit-To-Stand Test
  Score according to Rate of Perceived Exertion

CONTACTS AND LOCATIONS:
Locations (1):
- Papanikolaou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22556019/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39852605/